CLINICAL TRIAL: NCT02571569
Title: A Phase 1, First in Man, Multicenter, Open Label, Single Escalating Dose Study of BAY1093884 in Subjects With Severe Hemophilia Types A or B, With or Without Inhibitors
Brief Title: A Single Escalating Dose and Multiple Dose Study of BAY 1093884 in Subjects With Severe Hemophilia Types A or B, With or Without Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16144; 2014-003283-20 (EudraCT Number)
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Without inhibitors (Experimental): Dose escalation steps for participants without inhibitors - intravenous infusion and subcutaneous injection
  Interventions: Drug: BAY1093884
- With inhibitors (Experimental): Dose escalation steps for participants with inhibitors - intravenous infusion and subcutaneous injection
  Interventions: Drug: BAY1093884
- Without inhibitors_multiple dose (Experimental): Multiple dose cohort for participants without inhibitors - a single subcutaneous injection once a week for 6 weeks
  Interventions: Drug: BAY1093884

INTERVENTIONS:
Drug: BAY1093884 — Single escalating dose with a starting dose of 0.3 mg/kg for the first cohort. Drug will be administered via IV infusion over 1 hour and SC injection. Based on safety, PK and PD results the doses for the other cohorts will be determined.
  Arms: With inhibitors; Without inhibitors
Drug: BAY1093884 — Multiple dose cohort with a single 150-mg SC injection once a week for 6 weeks.
  Arms: Without inhibitors_multiple dose

SUMMARY:
Investigate the safety, tolerability and pharmacokinetics of BAY1093884 after Intravenous (IV) and subcutaneous (SC) administration of increasing single doses and SC administration of multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Males with severe congenital Hemophilia A or B defined as <1% FVIII or Factor IX (FIX) concentration by measurement at the time of screening or from reliable prior documentation
* For subjects in Cohorts I-IV, I-SC1 and I-SC2; If history of inhibitors is evident, inhibitor titer of ≥5 Bethesda Units (BU) at screening or prior to screening at any time from medical records.
* Age: 18 to 65 years of age at screening
* Body mass index (BMI): 18 to 29.9 kg/m²

Exclusion Criteria:

* Subjects with known bleeding disorders (such as von Willebrand factor [vWF] deficiency, FXI deficiency, platelet disorders, or known acquired or inherited thrombophilia etc.) other than congenital Hemophilia A or B with or without inhibitors
* History of angina pectoris or treatment for angina pectoris
* History of coronary and/or peripheral atherosclerotic disease, congestive heart failure, disseminated intravascular coagulopathy, or stage 2 hypertension defined as systolic blood pressure (SBP) ≥160 mmHg or diastolic blood pressure (DBP) ≥100 mmHg even if controlled
* History of thrombophlebitis, venous / arterial thromboembolic diseases (particularly deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction, cerebrovascular accident, ischemic heart disease, transient ischemic attack)
* Known or suspected hypersensitivity of the immune system, history of anaphylactic reaction, known (clinically relevant) allergies, non-allergic drug reactions, or multiple drug allergies

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Number of participants (single dose cohors) with adverse events as measure of safety and tolerability | Up to 56 days
  Adverse events including abnormal laboratory findings and local injection site reactions
Plasma levels of anti-BAY1093884 antibodies | Pre-dose, Day 14, 21,28, 43 and 56
Plasma concentration of BAY1093884 characterized by AUC(0-tlast) | Day 0 [pre-dose (within 1 hour), at the end of infusion or injection (=1hr), 2hrs, 4hrs, 8hrs], Days 1, 3, 5, 7, 14, 21, 28, 43, and 56 (for cohorts 3, 4 and I-SC2, S-2, S-3) after the start of infusion
  AUC from time 0 to the last data point > LLOQ (lower limit of quantitation)
Plasma concentration of BAY1093884 characterized by AUC(0-tlast)/D | Day 0 [pre-dose (within 1 hour), at the end of infusion or injection (=1hr), 2hrs, 4hrs, 8hrs], Days 1, 3, 5, 7, 14, 21, 28, 43, and 56 (for cohorts 3, 4 and I-SC2, S-2, S-3) after the start of infusion
  AUC(0-last) divided by dose
Plasma concentration of BAY1093884 characterized by Cmax | Day 0 [pre-dose (within 1 hour), at the end of infusion or injection (=1hr), 2hrs, 4hrs, 8hrs], Days 1, 3, 5, 7, 14, 21, 28, 43, and 56 (for cohorts 3, 4 and I-SC2, S-2, S-3) after the start of infusion
  Maximum observed drug concentration in measured matrix after single dose administration
Plasma concentration of BAY1093884 characterized by Cmax/D | Day 0 [pre-dose (within 1 hour), at the end of infusion or injection (=1hr), 2hrs, 4hrs, 8hrs], Days 1, 3, 5, 7, 14, 21, 28, 43, and 56 (for cohorts 3, 4 and I-SC2, S-2, S-3) after the start of infusion
  Cmax divided by dose

SECONDARY OUTCOMES:
Tissue factor pathway inhibitor (TFPI) activity | Up to 77 days
Number of participants (multiple dose cohort) with adverse events as a measure of safety and tolerability | Up to 77 days
  Adverse events including abnormal laboratory findings and local injection site reactions
Plasma levels of anti-BAY1093884 antibodies (multiple dose cohort) | Pre-dose, Day 14, 28, 49 and 77
Plasma concentration of BAY1093884 characterized by AUC(0-7d and AUC(0-tau) (multiple dose cohort) | Day 0 (prior to start of SC injection) and 8 hrs after start of SC injection, Days 1, 3, 5 and Days 7, and Day 35 (prior to start of SC injection) and 8 hrs after start of SC injection on Day 35; Days 36, 38, 40, 42
  AUC from time 0 to 7d after first and last dose (AUC(0-tau)
Plasma concentration of BAY1093884 characterized by AUC(0-7d/D and AUC(0-tau)/D after multiple dose | Day 0 (prior to start of SC injection) and 8 hrs after start of SC injection, Days 1, 3, 5 and Days 7, and Day 35 (prior to start of SC injection) and 8 hrs after start of SC injection on Day 35; Days 36, 38, 40, 42
  AUC(0-7d) after first dose and AUC(0-tau) after last dose divided by dose
Plasma concentration of BAY1093884 characterized by Cmax after first dose and last dose (Cmax,md) | Day 0 (prior to start of SC injection) and 8 hrs after start of SC injection, Days 1, 3, 5 and Days 7, and Day 35 (prior to start of SC injection) and 8 hrs after start of SC injection on Day 35; Days 36, 38, 40, 42
  maximum observed drug concentration in measured matrix after first and last dose
Plasma concentration of BAY1093884 characterized by Cmax/D after first dose and last dose (Cmax,md/D) | Day 0 (prior to start of SC injection) and 8 hrs after start of SC injection, Days 1, 3, 5 and Days 7, and Day 35 (prior to start of SC injection) and 8 hrs after start of SC injection on Day 35; Days 36, 38, 40, 42
  Cmax after first and last dose divided by dose
Accumulation of BAY 1093884 in plasma as defined by ratio for Cmax and AUC (after first and last dose) | Day 0 (prior to start of SC injection) and 8 hrs after start of SC injection, Days 1, 3, 5 and Days 7, and Day 35 (prior to start of SC injection) and 8 hrs after start of SC injection on Day 35; Days 36, 38, 40, 42
  Cmax after last dose divided by Cmax after first dose, AUC after last dose divided by AUC after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Germany (2):
  - Giessen, Hesse
  - Berlin
- Suginami, Tokyo, Japan
- Ukraine (2):
  - Kiev
  - Lviv
- United Kingdom (2):
  - London
  - Manchester